CLINICAL TRIAL: NCT00689481
Title: A Multicenter, Randomized, Double-Blind, Phase 3 Study of the Safety and Efficacy of Emulsion Formulation U0267 , Versus Vehicle Foam in Subjects With Plaque-type Psoriasis
Brief Title: Study to Compare U0267 Against Vehicle in Subjects With Plaque-type Psoriasis Two of Two Phase 3 Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114742; U0267-302 (Other: Stiefel)
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2010-12-08 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Psoriasis
Keywords: Plaque-type Psoriasis; psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- U0267 foam (Experimental): U0267 is a vitamin D3 analog (calcipotriene) foam. It is applied twice a day for 8 weeks to psoriasis lesions on the body.
  Interventions: Drug: U0267 Foam
- Vehicle foam (Placebo Comparator): Vehicle foam is the same as the U0267 foam except that it does not have the active ingredient. It is applied twice a day for 8 weeks to psoriasis lesions on the body.
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: U0267 Foam — All treatments will be administered topically twice daily (morning and evening) for 8 weeks to areas affected with psoriasis (excluding face and scalp).
  Arms: U0267 foam
Drug: Vehicle foam — All treatments will be administered topically twice daily (morning and evening) for 8 weeks to areas affected with psoriasis (excluding face and scalp).
  Arms: Vehicle foam

SUMMARY:
The purpose of the study is to demonstrate the safety and efficacy of U0267 in subjects with plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 12 years old and in good general health.
* Mild to moderate plaque-type psoriasis

Exclusion Criteria:

* Known allergy or other adverse reaction to calcipotriene or other vitamin D analogs; or to any component of the investigational formulations
* History of hypercalcemia or of vitamin D toxicity.
* Diagnosis of generalized pustular or erythrodermic exfoliative psoriasis.
* Other serious skin disorder or any chronic medical condition that is not well controlled.
* Use of non-biologic systemic anti-psoriatic therapy or biologic therapy within four weeks of enrollment.
* Use of topical therapies that have a known beneficial effect on psoriasis, within 2 weeks of enrollment.
* Systemic medications for other medical conditions that are known to affect psoriasis within the past four weeks of enrollment.
* Use of any investigational therapy within 4 weeks of enrollment.
* Pregnant women, women who are breast feeding, or sexually active women of child bearing potential who are not practicing an acceptable method of birth control.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (12):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Center for Dermatology Cosmetic and Laser Surgery, Fremont, California
  - Advanced Dermatology & Cosmetic Surgery, Ormond Beach, Florida
  - Adult & Pediatric Dermatology, Overland Park, Kansas
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - The Center for Dermatology at Lifetime Health, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Dermatology Consultants, Inc., Cincinnati, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - The Skin Wellness Center, PC, Knoxville, Tennessee
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Feldman SR, Matheson R, Bruce S, Grande K, Markowitz O, Kempers S, Brundage T, Wyres M; U0267-301 & 302 Study Investigators. Efficacy and safety of calcipotriene 0.005% foam for the treatment of plaque-type psoriasis: results of two multicenter, randomized, double-blind, vehicle-controlled, phase III clinical trials. Am J Clin Dermatol. 2012 Aug 1;13(4):261-71. doi: 10.2165/11630710-000000000-00000. PMID 22587791
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114742 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcipotriene Foam: Calcipotriene Foam is a vitamin D3 analog (calcipotriene) foam. It is applied twice a day for 8 weeks to psoriasis lesions on the body.
- Vehicle Foam: Vehicle foam is the same as the Calcipotriene Foam except that it does not have the active ingredient. It is applied twice a day for 8 weeks to psoriasis lesions on the body.
Period: Overall Study
Arm/Group | Calcipotriene Foam | Vehicle Foam
Started | 214 | 109
Completed | 190 | 95
Not Completed | 24 | 14
Not completed — Adverse Event | 7 | 1
Not completed — Lost to Follow-up | 4 | 3
Not completed — Lack of Efficacy | 4 | 3
Not completed — Non-compliance with study treatment | 1 | 1
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Excluded medication started during study | 0 | 1
Not completed — Subject early term, left on vacation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcipotriene Foam | Vehicle Foam | Total
Number analyzed (Participants) | 214 | 109 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (14.2) | 47.5 (16.9) | 47.8 (15.2)
Age, Customized [Number; unit: participants]
  12 to < 18 years | 2 | 3 | 5
  18 to < 65 years | 185 | 88 | 273
  > 65 years | 27 | 18 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 59 | 167
  Male | 106 | 50 | 156
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 3 | 13
  Black | 5 | 4 | 9
  Mulitracial | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 194 | 99 | 293
Disease Characteristic - Erythema [Number; unit: participants] — Disease characteristics of Erythema at baseline
  participants
    Light red coloration | 52 | 30 | 82
    Moderate red coloration | 158 | 76 | 234
    Bright red coloration | 4 | 3 | 7
Disease Characteristic - Scaling [Number; unit: participants] — Disease characteristics of Scaling at baseline
  participants
    Minimal | 1 | 0 | 1
    Mild | 65 | 33 | 98
    Moderate | 145 | 76 | 221
    Marked | 2 | 0 | 2
    Severe | 1 | 0 | 1
Disease Characteristic - Plaque Thickness [Number; unit: participants] — Disease characteristics of Plaque Thickness at baseline
  participants
    Possible but difficult to ascertain | 1 | 1 | 2
    Slight but definite elevation | 66 | 41 | 107
    Moderate elevation | 144 | 66 | 210
    Marked elevation | 2 | 1 | 3
    Very marked elevation | 1 | 0 | 1
Disease Characteristic - Target Lesion Location [Number; unit: participants] — Disease characteristics of Target Lesion Location at baseline
  participants
    Arm | 53 | 27 | 80
    Leg | 129 | 55 | 184
    Trunk | 32 | 27 | 59
Disease Characteristic - Investigator Static Global Assesssment (ISGA) [Number; unit: participants] — Disease characteristics of ISGA at baseline
  participants
    Mild | 56 | 31 | 87
    Moderate | 158 | 78 | 236
Disease Characteristic - Subject's Global Assessment [Number; unit: participants] — Disease characteristics of Subject's Global Assessment at baseline
  participants
    Almost clear | 2 | 2 | 4
    Mild | 18 | 9 | 27
    Moderate | 62 | 26 | 88
    Very noticeable | 96 | 55 | 151
    Severe | 36 | 17 | 53
Disease Characteristic - Percent BSA (extent of psoriasis) [Mean (Standard Deviation); unit: percentage] — Disease characteristics of Percent of BSA (extent of psoriasis) at baseline
  percentage | 6.3 (4.7) | 6.4 (5.2) | 6.4 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Success, Assessed Per the Investigator's Static Global Assessment
Description: Assessment (on a scale of 0 to 4) was made as a visual average of all lesions, except those on the face/scalp. 0=clear; minor residual discoloration; no erythema/scaling/plaque thickness (PT). 1=almost clear; occasional fine scale/faint erythema/barely perceptible PT. 2=mild; fine scales predominate; light red coloration/mild PT. 3=moderate; coarse scales predominate; moderate red coloration/moderate PT. 4=severe; thick tenacious scale predominates; deep red coloration/severe PT. Treatment success=ISGA score 0 or 1, and a minimum improvement in the ISGA score of 2 grades from BL to week 8.
Time Frame: 8 weeks
Population: Intent-to-Treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 214 | 109
participants | 58 | 17
Statistical Analysis 1: Comparison: Calcipotriene Foam vs Vehicle Foam; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel; Stratified by pooled center
Statistical Analysis 2: Comparison: Calcipotriene Foam vs Vehicle Foam; Consistency of results across investigative centers was verified using the Breslow-Day test of homogeneity the odds ration using a significance level of 0.1; Test type: Superiority or Other; p = 0.843, Breslow-Day test; Breslow-Day test of the homogeneity of the odds ratio using a 0.1 significance level

2. Secondary Outcome: Number of Subjects With a Target Lesion Score of 0 or 1 for Erythema and at Least a 2-grade Improvement From Baseline at Week 8
Description: Erythema was assessed on a 6-point scale. 0=no evidence of erythema; hyperpigmentation may be present. 1=faint erythema. 2=light red coloration. 3=moderate red coloration. 4=bright red coloration. 5=dusky to deep red coloration.
Time Frame: 8 Weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 214 | 109
participants | 67 | 22
Statistical Analysis 1: Comparison: Calcipotriene Foam vs Vehicle Foam; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel; Stratified by pooled center

3. Secondary Outcome: Number of Subjects With a Target Lesion Score of 0 or 1 for Scaling and at Least a 2-grade Improvement From Baseline at Week 8
Description: Scaling was assessed on a 6-point scale. 0=no evidence of scaling. 1=minimal; occasional fine scale over less than 5% of the lesion. 2=mild, fine scales predominate. 3=moderate; course scales predominate. 4=marked; thick non-tenacious scale predominates. 5=severe; very thick tenacious scale predominates.
Time Frame: 8 Weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 214 | 109
participants | 72 | 20
Statistical Analysis 1: Comparison: Calcipotriene Foam vs Vehicle Foam; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel — P-value is significant based on the Holm stepwise closed testing procedure to control multiplicity for the key secondary analyses if primary analysis was significant; Stratified by pooled center

4. Secondary Outcome: Number of Subjects With a Target Lesion Score of 0 for Plaque Thickness at Week 8
Description: Plaque thickness was assessed on a 6-point scale. 0=no evidence of plaque thickness. 1=barely perceptible plaque thickness, approximately 0.5 millimeters (mm). 2=mild plaque thickness, approximately 1 mm. 3=moderate plaque thickness, approximately 1.5 mm. 4=marked plaque thickness, approximately 2 mm. 5=severe plaque thickness, approximately 2.5 mm or more.
Time Frame: 8 Weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 214 | 109
participants | 42 | 12
Statistical Analysis 1: Comparison: Calcipotriene Foam vs Vehicle Foam; Test type: Superiority or Other; p = 0.052, Cochran-Mantel-Haenszel; Stratified by pooled center

5. Secondary Outcome: Number of Subjects Who Have an ISGA Score of 0 or 1 at Week 8
Description: Assessment (on a scale of 0 to 4) was made as a visual average of all lesions, except those on the face/scalp. 0=clear; minor residual discoloration; no erythema/scaling/plaque thickness (PT). 1=almost clear; occasional fine scale/faint erythema/barely perceptible PT. 2=mild; fine scales predominate; light red coloration/mild PT. 3=moderate; coarse scales predominate; moderate red coloration/moderate PT. 4=severe; thick tenacious scale predominates; deep red coloration/severe PT.
Time Frame: 8 Weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 214 | 109
participants | 78 | 27
Statistical Analysis 1: Comparison: Calcipotriene Foam vs Vehicle Foam; Test type: Superiority or Other; p = 0.033, Cochran-Mantel-Haenszel; Stratified by pooled center

6. Secondary Outcome: Number of Subjects Who Have Treatment Success at Week 8 Analyzed by Baseline ISGA (Mild or Moderate)
Description: as for outcome 1
Time Frame: 8 Weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Calcipotriene Foam | Vehicle Foam
Number analyzed (Participants) | 214 | 109
participants
  Mild | 8 | 4
  Moderate | 50 | 13
Statistical Analysis 1: Comparison: Calcipotriene Foam vs Vehicle Foam; Comparison of calcipotriene foam and vehicle foam for patients who had mild disease at baseline; Test type: Superiority or Other; p = 0.859, Cochran-Mantel-Haenszel; Stratified by pooled center
Statistical Analysis 2: Comparison: Calcipotriene Foam vs Vehicle Foam; Comparison of calcipotriene foam and vehicle foam for patients who had moderate disease at baseline; Test type: Superiority or Other; p = 0.015, Cochran-Mantel-Haenszel; Stratified by pooled center

ADVERSE EVENTS:
Arm/Group | Calcipotriene Foam | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 0/214 | 1/109
Other Adverse Events (participants affected / at risk) | 0/214 | 0/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcipotriene Foam (N=214) | Vehicle Foam (N=109)
Unilateral deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.